CLINICAL TRIAL: NCT02578329
Title: A Randomized Intervention Study to Assess the Effect of the Mediterranean Diet on the Plasma Fatty Acid Profile
Brief Title: An Intervention Study to Assess the Effect of the Mediterranean Diet on the Plasma Fatty Acid Profile
Acronym: RISMED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Principal Investigator, Fabrizio Veglia, Doctor, Centro Cardiologico Monzino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R194/14 - CCM203
Record Dates: First submitted 2015-07-23; First posted 2015-10-16 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Coronary Artery Disease
Keywords: Mediterranean diet; blood fatty acid; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Med Diet (Experimental): Intensively advised Mediterranean diet
  Interventions: Behavioral: Intensively advised Mediterranean diet
- Low Fat diet (Active Comparator): usual low-fat dietary advice
  Interventions: Behavioral: usual low-fat dietary advice

INTERVENTIONS:
Behavioral: Intensively advised Mediterranean diet — Mediterranean Diet: fatty fish 3 times/week; legumes 2-3 times/week; vegetables twice/day; fresh fruits twice/day; 30 to 45g olive oil/day; 1-2 glasses red wine/day; less than 150g red meat/week
  Arms: Med Diet
Behavioral: usual low-fat dietary advice — usual low-fat dietary advice for cardiovascular disease
  Arms: Low Fat diet

SUMMARY:
The purpose of this study is to determine whether a Mediterranean Diet, personalized in terms of total calories, total lipids and balanced in terms of saturated, mono- and poly-unsaturated lipids, corrects the adverse fatty acid profile of patients with CHD and reduces markers of oxidative stress and inflammation more effectively than a low-fat dietary advice.

DETAILED DESCRIPTION:
Geographical differences in the incidence of CardioVascular Disease (CVD) show a lower risk in countries of south Europe compared with north and east Europe and USA. The Mediterranean Diet (MD) has been the most frequently invoked factor to explain these differences, but the underlying mechanisms are still unclear. On the other hand, blood fatty acid (FA) composition has been shown to be strongly related to cardiovascular risk, presumably through changes in oxidative stress and inflammatory pathways, two mechanisms involved in the pathogenesis of atherothrombosis. Preliminary data from our group suggest that patients with Coronary Heart Disease (CHD) adhere less to features of MD and exhibit a different fatty acid profile compared to healthy subjects. We speculate that MD may reduce oxidative stress and inflammatory markers, and reverse the unfavorable blood fatty acid profile observed in patients with CHD. Even though single MD components (wine, olive oil, vegetables, fish, etc) have shown beneficial effects on oxidative stress, inflammation and CardioVascular (CV) risk, evidence indicates that these effects are mostly related to the extent of compliance with the whole MD, which comprises possible synergism between food components. For this reason, the present study will consider the whole MD and not single components.

Design: randomized, parallel groups, open-label, intervention trial. Intervention: an intensively advised MD (fatty fish at least 3 times/week; legumes 2-3 times/ week; vegetables twice a day; fruits twice/day; 30-45g olive oil/day; 1-2 glasses of red wine/day, not more than 150g red meat/week), personalized in terms of calories, total lipids and balanced in terms of saturated, mono- and poly-unsaturated lipids (n= 75) vs. usual low-fat dietary advice (n=75) for 3 months. Participants: males and females, age 30-75, with a recent history of coronary revascularization, randomized after clinical stabilization (at least 60 days after any coronary procedure or event).

At baseline and after intervention in both groups:

Dietary assessment: using the EPIC questionnaire, a well validated dietary recall tool.

Blood, urinary and fecal samples: routine biochemical determinations, blood fatty acid composition by gas-chromatography, C reactive protein and oxidative stress markers (urinary isoprostanes, whole blood reduced and oxidized glutathione by Liquid Chromatography- Mass Spectrometry (LC-MS/MS), plasma alpha- and gamma-tocopherol by High Performance Liquid Chromatography (HPLC) with fluorimetric detector), gene expression and/or epigenome in peripheral whole blood cells (as an index of global changes of inflammation/immune response), intestinal microbiome.

Statistical analysis: Principal component analysis to characterize fatty acid patterns. Score of Trichopoulou to assess adherence to MD.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of coronary artery disease
* recent history of a first coronary revascularization
* at least 60 days after any coronary procedure or event
* age between 30 and 75 years

Exclusion Criteria:

* diagnosis of diabetes mellitus
* food intolerance to any component of the mediterranean diet
* BMI < 19 or > 33
* assuming drugs or food supplements with omega-3 fatty acids or natural or synthetic antioxidants.
* patients already adherent to a full mediterranean diet

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-10 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Change of whole blood fatty acid profile | three months
  Urinary isoprostanes (8-iso-PGF2-alpha will be measured at randomization and after dietary intervention by liquid chromatography-tandem mass spectrometry (LC-MS/MS) methods.

SECONDARY OUTCOMES:
Effect of Mediterranean diet on urinary isoprostanes | three months
  Urinary isoprostanes (8-iso-PGF2-alpha will be measured at randomization and after dietary intervention by liquid chromatography-tandem mass spectrometry (LC-MS/MS) methods.
Effect of Mediterranean diet on oxidized glutathione | three months
  Whole blood oxidized glutathione (GSSG) will be measured at randomization and after dietary intervention by liquid chromatography-tandem mass spectrometry (LC-MS/MS) methods.
Effect of Mediterranean diet on reduced glutathione | three months
  Whole blood reduced glutathione (GSH) will be measured at randomization and after dietary intervention by liquid chromatography-tandem mass spectrometry (LC-MS/MS) methods.
Effect of Mediterranean diet on plasma Vitamin E | three months
  Plasma vitamin E (alpha- and gamma-tocopherol) will be measured at randomization and at the end of the study by liquid chromatography-tandem mass spectrometry (LC-MS/MS) methods.
Effect of Mediterranean diet on Low-grade systemic inflammatory status | three months
  Effect of Mediterranean diet on Low-grade systemic inflammatory status will be assessed at randomization and at the end of the study by high sensitivity C-Reactive protein (hs-CRP) measured by immunoturbidimetry
Effect of Mediterranean diet on peripheral blood transcriptome | three months
  Whole transcriptome analysis will be performed by next-generation sequencing (NGS) on whole-blood derived RNA at randomization and after dietary intervention. Comparisons will be made between the two groups (MD vs. control diet). The outcome measure will be significant differential expression (fold-change) both at gene and gene-set levels.
Significant differences in the relative abundance of the operational taxonomic units (OTU) within subjects | three months
  Changes in gut bacterial composition (microbiome) will be assessed by massive parallel sequencing of the hypervariable regions of the 16S (Svedberg) rRNA (ribosomal ribonucleic acid) gene on genomic DNA isolated from stool samples at the three time-points, in order to identify the intestinal bacterial phylotypes. The outcome measure will be significant differences in the relative abundance of the operational taxonomic units (OTU) within subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Cardiologico Monzino, IRCCS, Milan, MI, Italy